CLINICAL TRIAL: NCT02757885
Title: Transplantation Using Reduced Intensity Approach for Patients With Sickle Cell Disease From Mismatched Family Donors of Bone Marrow
Brief Title: Transplantation for Patients With Sickle Cell Disease From Mismatched Family Donors of Bone Marrow
Acronym: TRANSFORM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Suhag Parikh, Professor of Pediatrics, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00080955
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Sickle Cell Disease
Keywords: bone marrow transplant
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Bone Marrow Transplantation; Hydroxyurea; Thiotepa; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bone Marrow Recipient (Experimental): Single arm open label study: Participants with sickle cell disease (SCD) will receive bone marrow from a human leukocyte antigen (HLA) mismatched donor.
  Interventions: Procedure: Bone Marrow Transplant (BMT); Drug: Hydroxyurea; Drug: Thiotepa; Drug: Fludarabine monophosphate; Drug: Cyclophosphamide; Other: Rabbit Anti-thymocyte Globulin; Radiation: Total Body Irradiation

INTERVENTIONS:
Procedure: Bone Marrow Transplant (BMT) — Participants will receive a bone marrow infusion from a human leukocyte antigen (HLA) mismatched donor through a central venous catheter.
Drug: Hydroxyurea — Hydroxyurea is part of the bone marrow transplant preparative regimen. Hydroxyurea will be administered at a dose of 30 mg/kg orally as a single daily dose for 90 days (from day -100 to day-10). Hydroxyurea dosing will be based on adjusted body weight in participants weighing >125% ideal body weight.
Drug: Thiotepa — Thiotepa is part of the bone marrow transplant preparative regimen. Thiotepa will be administered at a dose of 10mg/kg intravenously (IV) over 2 hours or per institutional guidelines on day -7. Thiotepa dosing will be based on adjusted body weight in patients weighing >125% ideal body weight.
Drug: Fludarabine monophosphate — Fludarabine is part of the bone marrow transplant preparative regimen. Fludarabine 30 mg/m2/day will be administered from day -7 to day -3 (for a total of 150 mg/m2 over 5 consecutive days) and administered intravenously (IV) over a minimum of 30 minutes. In participants weighing > 125% ideal body weight, fludarabine will be dose based upon adjusted body weight.
Drug: Cyclophosphamide — Cyclophosphamide is part of the bone marrow transplant preparative regimen. Cyclophosphamide will be administered on days -6 and -5 prior to bone marrow infusion at a dose of 14.5 mg/kg intravenously (IV) infused over 1-2 hours.
  Post bone marrow infusion cyclophosphamide will be infused on days +3 (between 60 and 72 hours post marrow infusion) and +4 (approximately 24 hours after day +3 dose) at a dose of 50 mg/kg IV infused over 1-2 hours.
  For participants weighing more than 125% of their ideal body weight, dosing will be based on adjusted ideal body weight.
Other: Rabbit Anti-thymocyte Globulin — Rabbit anti-thymocyte globulin (ATG) is part of the bone marrow transplant preparative regimen. It is an infusion of rabbit-derived antibodies against human T cells used for prevention of acute rejection in organ transplantation. Rabbit ATG will be administered on day -9 at 0.5 mg/kg and on days -8 and -7 at 2 mg/kg (for a total dose 4.5 mg/kg).
Radiation: Total Body Irradiation — Participants will receive 200 cGy of TBI in a single fraction.

SUMMARY:
The purpose of this study is to learn if it is possible and safe to treat persons with severe sickle cell disease (SCD) by bone marrow transplant (BMT) from human leukocyte antigen (HLA) half-matched related donors. Preparation before transplant includes the chemotherapy drugs hydroxyurea, fludarabine, thiotepa, anti-thymocyte globulin, and cyclophosphamide. It also includes radiation.

DETAILED DESCRIPTION:
The purpose of this study is to learn if it is possible and safe to treat persons with severe sickle cell disease (SCD) by bone marrow transplant (BMT) from human leukocyte antigen (HLA) half-matched related donors. Preparation before transplant includes the chemotherapy drugs hydroxyurea, fludarabine, thiotepa, anti-thymocyte globulin, and cyclophosphamide. It also includes radiation.

Investigators also seek to understand the side effects of BMT in adolescents and young adults with SCD and measure how often serious side effects occur including those that are expected and unexpected. After transplant, investigators will measure the health of the body organs that ordinarily would have been damaged by having SCD in addition to testing the lungs, brain, and kidneys.

ELIGIBILITY:
Inclusion Criteria:

1. Disease severity: Participants with SCD who have 1 or more of the following (i-v).

   * Clinically significant neurologic event (stroke) or any neurological deficit lasting > 24 hours;
   * History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea);
   * History of three or more severe pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea);
   * Administration of regular red blood cell (RBC) transfusion therapy, defined as receiving 8 or more transfusions per year for ≥ 1 year to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and ACS). Patients on chronic transfusion who have to discontinue transfusion because of allo-sensitization will be eligible.
   * An echocardiographic finding of tricuspid valve regurgitant jet (TRJ) velocity ≥ 2.7 m/sec. Patients under the age of 18 years must have cardiac catheterization proven pulmonary arterial hypertension to qualify on this eligibility criterion.
2. Age: Patients must be 15 - 40 years of age inclusive OR if younger than 15 years must be pubertal
3. Adequate physical function as measured by:

   * Karnofsky/Lansky performance score ≥ 60
   * Cardiac function: Left ventricular ejection fraction (LVEF) > 40% or LV shortening fraction > 26% by cardiac echocardiogram or by MUGA scan.
   * Pulmonary function: Pulse oximetry with a baseline O2 saturation of ≥ 85% and DLCO > 40% (corrected for hemoglobin).
   * Renal function: Serum creatinine ≤ 1.5 x the upper limit of normal for age as per local laboratory and 24 hour urine creatinine clearance > 70 mL/min/1.73 m2 or GFR > 70 mL/min/1.73 m2 by radionuclide GFR.
   * Hepatic function: Serum conjugated (direct) bilirubin < 2 x upper limit of normal for age as per local laboratory and ALT and AST < 5 x upper limit of normal as per local laboratory. Patients with hyperbilirubinemia as a consequence of hyperhemolysis, or who experience a sudden, profound change in the serum hemoglobin after a RBC transfusion, are not excluded.
   * For participants with a suitable donor who meet eligibility criteria and are willing to proceed to HCT, if they have received chronic transfusion therapy for ≥ 1 year and have clinical evidence of iron overload by serum ferritin or MRI, an evaluation by liver biopsy is required. Histological examination of the liver must document the absence of cirrhosis, bridging fibrosis, and active hepatitis. The absence of bridging fibrosis will be determined using the histological grading and staging scale
4. Suitable Donor: To undergo transplantation on this study, participants must have an adult first degree relative who shares at least 1 human leukocyte antigen (HLA) haplotype with the participant, does not have SCD or other hemoglobinopathy, and is in good health; if these criteria are met, they will be allowed to serve as donors. Relatives with sickle cell trait are not excluded as donors. When more than 1 donor is available, the donor with the fewest HLA allele mismatches will be chosen, unless the patient had donor anti-HLA antibodies or there was a medical reason to exclude the donor. If donor anti-HLA antibodies are detected, the next best related match will be chosen. Umbilical cord blood or peripheral blood stem cell donors will not be accepted.

Exclusion Criteria:

* Availability of HLA matched sibling or 8 of 8 HLA-A, B, C and DRB1 matched unrelated donor
* Presence of donor specific antibodies in the patient
* Histological examination of the liver must document the absence of cirrhosis, bridging fibrosis and active hepatitis. The absence of bridging fibrosis will be determined using the histological grading and staging scale as described by Ishak and colleagues (1995). The presence of bridging fibrosis will be an exclusion criterion.
* Uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment
* Seropositivity for HIV
* Previous hematopoietic cell transplantation (HCT)
* Participation in a clinical trial in which the patient received an investigational drug or device or off-label use of a drug or device within 3 months of enrollment
* Demonstrated lack of compliance with prior medical care
* Unwilling to use approved contraception for at least 6 months after transplant
* A history of substance abuse in the last 5 years that interferes with care
* Pregnant or breast-feeding females at the time of consideration for HCT

Donor Selection Criteria:

Preference will be given to related marrow donors who are 2-4 (out of 8) HLA antigen mismatched and towards whom the recipient does not have donor specific antibodies. Donors will sign an informed consent disclosing that the marrow donation will be used by a patient participating in this study. The donor must be matched with the recipient for at least 4 of 8 HLA alleles (HLA -A, -B, -C and -DRB1 by allele-level DNA methodology). The target total nucleated cell count (TNC) is 3.5-8.0 x 108/kg of recipient weight. Marrow will be collected without mobilization. Mobilized peripheral blood stem cell (HPC-A) collections will not be permitted. Donors must undergo hemoglobinopathy screening by electrophoresis; donors who have a hemoglobinopathy will be excluded but trait condition is acceptable.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta (CHOA) in Atlanta, Georgia, USA. Participant enrollment began July 10, 2019, and all follow up was complete by December 14, 2021.
Pre-assignment Details: Donors in this trial were not considered research participants. Donors were consented per standard of care; these consents were obtained by non-research physicians. Demographics and/or other outcomes were not collected on the donors. Donor selection criteria are included in the protocol to specify the donor preference to be studied in this particular transplant recipient group. Donors provided consent disclosing that the marrow donation would be used by a recipient who was in a research study.
Groups:
- Bone Marrow Recipient: Patients with SCD will receive a Bone Marrow Transplant (BMT) infusion from an HLA-mismatched donor through a central venous catheter.
  Hydroxyurea (HU): HU is part of the BMT preparative regimen. Dose: 30 mg/kg orally once a day for 90 days (days -100 to -10). HU Dose adjusted in patients weighing >125% IBW.
  Thiotepa: Thiotepa is part of the BMT preparative regimen. Dosed at 10mg/kg intravenously (IV) over 2 hrs or per institutional guidelines on day -7. Dose adjusted in patients weighing >125% IBW.
  Fludarabine (FCR) monophosphate: FCR is part of the BMT preparative regimen. FCR given IV: 30 mg/m2/day over a min. of 30 minutes on days -7 to -3 (150 mg/m2 over 5 consecutive days). Dose adjusted in patients weighing >125% IBW.
  Cyclophosphamide (CP): CP is part of the BMT preparative regimen. Given over 1-2 hrs on days -6 and -5 prior to BMT infusion at a dose of 14.5 mg/kg IV.
  Post BMT infusion CP is infused over 1-2 hrs on days +3 (60- and 72-hrs post BMT infusion) and +4 (approx. 24 hrs after day +3 dose) at a dose of 50 mg/kg IV. Dose adjusted in patients weighing >125% IBW.
  Rabbit Anti-thymocyte Globulin (ATG): Rabbit (ATG) is part of the BMT preparative regimen, an infusion of rabbit-derived antibodies against human T cells used for the prevention of acute rejection in organ transplantation. Rabbit ATG is given on days -9 at 0.5 mg/kg and on days -8 and -7 at 2 mg/kg (4.5 mg/kg).
  Total Body Irradiation: Participants will receive 200 cGy of TBI in a single fraction.
Period: Overall Study
Arm/Group | Bone Marrow Recipient
Started | 10
Completed | 6
Not Completed | 4
Not completed — Screen Failures | 4

BASELINE CHARACTERISTICS:
Groups:
- Bone Marrow Recipient: Patients with SCD will receive a Bone Marrow Transplant (BMT) infusion from an HLA-matched donor through a central venous catheter.
  Hydroxyurea (HU): HU is part of the BMT preparative regimen. Dose: 30 mg/kg orally once a day for 90 days (days -100 to -10). HU Dose adjusted in patients weighing >125% IBW.
  Thiotepa: Thiotepa is part of the BMT preparative regimen. Dosed at 10mg/kg intravenously (IV) over 2 hrs or per institutional guidelines on day -7. Dose adjusted in patients weighing >125% IBW.
  Fludarabine (FCR) monophosphate: FCR is part of the BMT preparative regimen. FCR given IV: 30 mg/m2/day over a min. of 30 minutes on days -7 to -3 (150 mg/m2 over 5 consecutive days). Dose adjusted in patients weighing >125% IBW.
  Cyclophosphamide (CP): CP is part of the BMT preparative regimen. Given over 1-2 hrs on days -6 and -5 prior to BMT infusion at a dose of 14.5 mg/kg IV.
  Post BMT infusion CP is infused over 1-2 hrs on days +3 (60- and 72-hrs post BMT infusion) and +4 (approx. 24 hrs after day +3 dose) at a dose of 50 mg/kg IV. Dose adjusted in patients weighing >125% IBW.
  Rabbit Anti-thymocyte Globulin (ATG): Rabbit (ATG) is part of the BMT preparative regimen, an infusion of rabbit-derived antibodies against human T cells used for the prevention of acute rejection in organ transplantation. Rabbit ATG is given on days -9 at 0.5 mg/kg and on days -8 and -7 at 2 mg/kg (4.5 mg/kg).
  Total Body Irradiation: Participants will receive 200 cGy of TBI in a single fraction.
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Rate
Description: Event-free Survival (EFS) is defined as the survival with stable donor erythropoiesis with no new clinical evidence of sickle cell disease (SCD). Primary or late graft rejection with disease recurrence or death will count as events for this endpoint.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 5

2. Primary Outcome: Primary Graft Rejection Rate
Description: Primary graft rejection is defined as the absence of donor cells assessed by peripheral blood chimerism assays on day 42. Primary graft rejection can be accompanied by pancytopenia and marrow aplasia or by autologous hematopoietic reconstitution without aplasia.
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 1

3. Primary Outcome: Late Graft Rejection Rate
Description: The absence of donor hematopoietic cells in peripheral blood beyond day 42 up to 1 year in a patient who had initial evidence of hematopoietic recovery with > 20% donor cells will be considered a late graft rejection.
Time Frame: Day 42 Post transplant up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 0

4. Primary Outcome: Rate of Disease Recurrence
Description: Disease recurrence is defined as the return of sickle erythropoiesis (HbS level > 70%) and the absence of donor cell representation.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 1

5. Secondary Outcome: Overall Survival Rate
Description: Overall survival is defined as survival with or without sickle cell disease (SCD) after hematopoietic cell transplantation (HCT).
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 6

6. Secondary Outcome: Cumulative Incidence of Neutrophil Engraftment and Platelet Engraftment.
Description: Cumulative incidence of Neutrophil Engraftment and Platelet Engraftment. Neutrophil engraftment is defined as the first of 3 measurements on different days when the patient has an absolute neutrophil count of ≥ 500/µL after conditioning.
  Platelet engraftment is defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/µL and did not receive a platelet transfusion in the previous 7 days.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 5

7. Secondary Outcome: Chimerism Rate Following Hematopoietic Cell Transplantation for Sickle Cell Disease
Description: Genomic DNA extracted from peripheral blood will be analyzed for variable number of tandem repeats (VNTR) to detect donor engraftment in myeloid and lymphoid fractions.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 5

8. Secondary Outcome: Frequency of Idiopathic Pneumonia Syndrome (IPS)
Description: IPS is diagnosed by evidence of widespread alveolar injury:
  1. Radiographic evidence of bilateral, multi-lobar infiltrates (by chest x-ray or CT scan); AND
  2. Evidence of abnormal respiratory physiology based upon oxygen saturation (SpO2) < 93% on room air or the need for supplemental oxygen to maintain oxygen saturation ≥ 93%; AND
  3. Absence of active lower respiratory tract infection
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 0

9. Secondary Outcome: Veno-occlusive Disease (VOD) Rate
Description: VOD is diagnosed by the presence of ≥ 2 of the following with no other identifiable cause for liver disease:
  1. Jaundice (direct bilirubin ≥ 2 mg/dL or > 34 μmol/L)
  2. Hepatomegaly with right upper quadrant pain
  3. Ascites and/or weight gain (> 5% over baseline)
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 0

10. Secondary Outcome: Rate of Central Nervous System (CNS) Toxicity
Description: CNS toxicity will be defined as seizures, CNS hemorrhage, or PRES. PRES is defined as an increased diffusion coefficient in areas of T2 hyperintensity on diffusion-weighted imaging in the context of clinical symptoms or physical findings including headache, seizures, visual disturbances, and altered level of consciousness.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 2

11. Secondary Outcome: Infection Rate
Description: Significant infections will be recorded including but not limited to bacterial or fungal sepsis, CMV reactivation with/without clinical disease, adenovirus infection, EBV PTLD, other significant viral reactivations or community-acquired viral infections and invasive mold infections.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 5

12. Secondary Outcome: Frequency of Stroke
Description: An overt stroke is defined as a focal neurologic event and neurologic deficit lasting > 24 hours with neuroimaging changes.
Time Frame: Up to One Year
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Recipient
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: Data collected up to one year post-transplant.
Arm/Group | Bone Marrow Recipient
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone Marrow Recipient (N=6)
Non-engraftment (Blood and lymphatic system disorders) | 1 (1) — Graft failure happens when the new cells don't make the new white blood cells, red blood cells, and platelets you need. This is also called "failure to engraft" or "non-engraftment.
Central Nervous System Toxicity (Nervous system disorders) | 2 (2) — Posterior reversible encephalopathy syndrome
Graft-versus-host disease (GVHD) (Immune system disorders) | 4 (9)
Thrombotic microangiopathy (TMA) (Blood and lymphatic system disorders) | 1 (1)
Epstein-Barr virus (EBV) (Infections and infestations) | 3 (4)
Deep vein thrombosis (DVT) (Blood and lymphatic system disorders) | 1 (1)
Cytomegalovirus infection (CMV) (Infections and infestations) | 1 (1)
BK virus (BKV) (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 4 (9)
Bacteriemia (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02757885/Prot_SAP_000.pdf